CLINICAL TRIAL: NCT04070495
Title: A Drug Interaction Study of KW-6356 and Clarithromycin or Rifampicin (A Drug Interaction Study With a CYP3A4/5 Inhibitor or Inducer)
Brief Title: A Drug Interaction Study of KW-6356 and Clarithromycin or Rifampicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6356-008
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Clarithromycin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clarithromycin (Experimental)
  Interventions: Drug: KW-6356; Drug: Clarithromycin
- Rifampicin (Experimental)
  Interventions: Drug: KW-6356; Drug: Rifampicin

INTERVENTIONS:
Drug: KW-6356 — A single oral dose will be administered at Day 1 and 15
Drug: Clarithromycin — 400mg, oral tablet (2 x 200mg), twice daily (BID), Day 8-28
  Arms: Clarithromycin
Drug: Rifampicin — 600mg, oral tablet (4 x 150mg), once daily (QD), Day 8-21
  Arms: Rifampicin

SUMMARY:
The purpose of this study is to investigate the effects of CYP3A4/5 inhibitor or inducer on the pharmacokinetics of KW-6356 when CYP3A4/5 inhibitor or inducer is orally administered to healthy Japanese men for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects having issued written consent to this study at their own discretion
2. Japanese men aged 20 to 44 years at the time of informed consent
3. Subjects with BMI ≥18.5 and <25.0 at screening
4. Subjects with screening results of; resting pulse rate: 40 to 100 bpm, systolic blood pressure: 90 to 139 mmHg, diastolic blood pressure: 40 to 89 mmHg

Exclusion Criteria:

1. Subjects with any current disease requiring treatment
2. Subjects having drug allergy or its history
3. Subjects having psychiatric disease or its history
4. Positive results for any of the following infection-related items examined at screening: hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, human T-lymphotropic virus (HTLV)-1 antibody, rapid plasma reagin (PRP) test, or Treponema pallidum (TP) antibody.
5. Subjects with clinically significant abnormality detected on 12-lead electrocardiogram (ECG) recorded prior to the first administration of investigational product.
6. Subjects categorized as patients listed in the warnings or contraindications section of the package insert of the perpetrator drug.
7. Subjects having used any drug (including over-the-counter [OTC] drugs, topical agents, vitamin preparations, health supplements, and Chinese herbal medicines) within 2 weeks prior to the first administration of investigational product.
8. Subjects having consumed grapefruit (including any food or beverage containing grapefruit) or any food or beverage containing St John's wort within 1 week prior to the first administration of investigational product.
9. Subjects having smoked or used smoking cessation agents (including chewing or eating of nicotine-containing products and application of nicotine patches) within 4 weeks prior to the first administration of investigational product.
10. Subjects having received inpatient treatment or surgery within 12 weeks prior to the first administration of investigational product.
11. Subjects having participated in a clinical study of a pharmaceutical product or a medical device or any equivalent study and used the investigational product or the unapproved medical device within 4 months prior to the first administration of investigational product.
12. Subjects having undergone ≥400 mL of blood collection within 12 weeks prior to the first administration of investigational product or ≥200 mL of blood collection within 4 weeks prior to the first administration of investigational product (for blood donation or clinical trial, etc.) or pheresis donation (plateletpheresis or plasmapheresis donation) within 2 weeks prior to the first administration of investigational product.
13. Subjects having issued no consent to adoption of any appropriate contraceptive method during the period from day of admission to 12 weeks after the final administration of the perpetrator drug. The appropriate contraceptive method is defined as sexual abstinence or use of 2 of the following contraceptive devices: condom, oral contraceptives, intrauterine device, and pessary.
14. Subjects having received KW-6356 before.
15. Other subjects unsuitable for participating in the study in the opinion of the investigator or subinvestigator.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratio of the pharmacokinetic parameter (AUC0-t) of KW-6356 in combination with or without a perpetrator drug | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.

SECONDARY OUTCOMES:
Geometric mean ratio of the major pharmacokinetic parameters (Cmax) of KW-6356 in combination with or without a perpetrator drug | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Geometric mean ratio of the major pharmacokinetic parameters (AUC0-∞) of KW-6356 in combination with or without a perpetrator drug | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Pharmacokinetic parameters (tmax) of KW-6356 | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Pharmacokinetic parameters (CL/F) of KW-6356 | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Pharmacokinetic parameters (Vz/F) of KW-6356 | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Pharmacokinetic parameters (t1/2) of KW-6356 | Starting just before intake of KW-6356 and continued until 168 or 336 hours after intake of KW-6356.
Plasma concentrations of a perpetrator drug | Starting just before intake of a perpetrator drug at Day 8 and continued until 12 or 24 hours after the last dose of a perpetrator drug.
Incidence of treatment-emergent adverse events | Starting 24 hours before intake of KW-6356 and continued until 14 days after the last dose of a perpetrator drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Co. LTA Sumida Hospital, Sumida-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided